CLINICAL TRIAL: NCT05128526
Title: Effect of Respiratory Combined Short Foot Exercises on Foot and Ankle Muscle Activity in Individuals With Pes Planus
Brief Title: Short Foot Exercises With Respiratuar Exercises
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Tezel Yıldırım Şahan, Clinical Researcher, Hacettepe University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: 2021/366
Record Dates: First submitted 2021-10-28; First posted 2021-11-22 (Actual); Last update posted 2022-11-29 (Actual); Status verified 2022-11

CONDITIONS: Exercise; Flatfoot
Keywords: pes planus; respiratory; exercise; short foot exercise
MeSH Terms: conditions — Motor Activity; Flatfoot | interventions — Exercise; Respiratory Rate

STUDY DESIGN:
Intervention Model Description: Two-way repeated analyses of variance were used to determine the statistical significance of muscles electromyography activity
Who Masked: Participant
Masking Description: Two-way repeated analyses of variance were used to determine the statistical significance of muscles electromyography activity
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Short foot exercise without respiratory exercises (Experimental): The participant will place by the researcher in the standing position so that the width between both feet will equal the width of the pelvis and the second toe will align with the patella. During the Short Foot Exercise, the participant will ask to position the spine straight, maintain the pelvis in a neutral position, and place the centerline of the body. The starting position will be set by the researcher under the same conditions as the midway between the feet. The subjects will give feedback from the researchers to assist in the maintenance of accurate body alignment. SFE, only in a standing position.
  The participants will keep in contact with the fibular head of the target bar to maintain a constant position during Short Foot Exercises. Afterward, surface EMG measurements will be taken from the same muscle groups for 10 seconds during the foot shortening exercises while without breathing.
  Interventions: Behavioral: exercise
- Short Foot Exercise With Respiratory Exercise (Experimental): The participants will keep in contact with the fibular head of the target bar to maintain a constant position during Short Foot Exercises. Afterward, surface EMG measurements will be taken from the same muscle groups for 10 seconds during the foot shortening exercises while with breathing.
  Interventions: Behavioral: respiratory

INTERVENTIONS:
Behavioral: exercise — Short foot exercises without respiratory exercises
  Other Names: short foot exercise
  Arms: Short foot exercise without respiratory exercises
Behavioral: respiratory — Short foot exercises with respiratory exercises
  Other Names: Short foot exercise
  Arms: Short Foot Exercise With Respiratory Exercise

SUMMARY:
Pes planus is a common foot problem since childhood, which may include loss of height of the medial longitudinal arch, which is the most important arch supporting the foot, valgus of the hindfoot, and abduction of the midfoot relative to the hindfoot. Muscle shortness, increased joint laxity with obesity, W-shaped sitting, male gender and genetic background are among the factors that can increase the incidence and severity of pes planus in the pediatric population. It has been shown in different studies that pes planus is carried into adulthood at a rate of 4-23%. It is known that there is oxygen consumption from the body during muscle contraction. For this reason, it has been shown in the literature that muscle oxygenation is better and the performance of the individual is better in exercises combined with breathing exercises in the exercise program. Therefore, the investigators hypothesized whether foot shortening exercises combined with breathing would have an effect on muscular activation during foot shortening exercises. It is seen that there is a limited number of studies in the literature evaluating the effect of breathing exercises and combined foot exercises on the activation of the muscles around the feet. For this reason, the aim of this study is to examine the effect of combined respiratory foot shortening exercises on the muscular activations of the foot circumference in individuals with flat feet. Two-way repeated analyses of variance will use to determine the statistical significance of Abductor Hallucis Longus, Tibialis Anterior, and Peroneus Longus electromyography activity. Participants: Ten participants with pes planus.The participants will perform Short Foot Exercises with and without respiratory exercises in sitting and standing positions. Main Outcome Measures: Surface electromyography will use to measure the activity of the Abductor Hallucis Longus, Tibialis anterior, Peroneus Longus. Respiratory exercises may be an effective method for reducing compensatory Tibialis Anterior activity and increasing Abductor Hallucis Longus muscle activity during Short Foot Exercises for individuals with pes planus.

DETAILED DESCRIPTION:
Ten volunteer individuals with flat feet, studying at the Faculty of Health Sciences, will be included in the study. The feet of the individuals who want to be included in the study will be examined by the researchers with the Navicular drop test. Individuals' age, height, weight, gender, shoe size will be questioned. Flat feet of individuals will be determined by the Navicular Drop test. The navicular drop test is a test used to measure the amount of pronation in the foot, which is obtained by subtracting the navicular height measured while standing with weight on the foot, from the navicular height measured in the sitting position without placing weight on the foot. While individuals are sitting on a chair with bare feet, the navicular tubercle will be marked on both feet and marked at the level of the navicular tubercle on a card on the floor. Afterward, the individual was asked to stand up, and the navicular tubercle alignment would be re-marked on the same card while giving full weight to the foot. The expression in mm of the distance between both lines will be recorded as the amount of navicular drop. The amount of navicular drop between 6 and 9 mm will be considered as normal Medial Longitudinal Arch, and if it is 10 mm or more, it will be considered as pes planus. Individuals will be divided into two groups according to the Navicular drop test. This research will consist of two groups, one group of individuals with flat feet and one group of individuals without flat feet. In both groups, foot shortening exercises will be applied in two different situations. The first case is the activation of the foot circumference muscles during the foot shortening exercises, and the second situation is the activation of the foot circumference muscles during the combination of the foot shortening exercises with the breathing exercises. Foot shortening exercise, in this exercise that works the small intrinsic muscles of the foot in isolation, the subjects will be asked to raise the medial foot and hold it in this position for 5 seconds while sitting on the ground with the feet in the subtalar neutral position, trying to bring the heel and fingers closer to each other. During the movement, the fingers will be warned not to bend participants' fingers to avoid a contraction in the long flexor muscles, while Participants will be asked to do 3 repetitions. After the individuals are given 5 minutes to rest the participants' feet, participants will be asked to combine the same exercise with breathing exercises. When the exercise is terminated, the situation will be returned to the start position. Muscular activations of the Tibialis anterior, Abductor Hallucis, and Peroneus Longus muscles will be measured with superficial kinesiological electromyography (EMG) device. The electrode sites will be prepared for the EMG signal by shaving and cleaning the skin with cotton dipped in alcohol to minimize output impedance and allow proper electrode bonding. Disposable Ag/AgCl superficial electrodes will be placed approximately 2 cm apart in the direction of the muscle fibers. Electrodes will be placed parallel to the muscle fibers at points recommended by Surface ElectroMyoGraphy for the Non-Invasive Assessments of Muscles (SENIAM). A detailed description of the electrode placements is as follows:

EMG electrodes for Abductor Hallucis will be attached from the anterior edge of the medial malleolus approximately 1-2 cm posterior to the navicular tuberosity, located just in front of the vertical line. For the Tibialis Anterior, the electrodes will be placed in the area corresponding to the one-third between the tip of the head of the fibula and the medial malleolus. For the Peroneus Longus muscle, the electrodes will be placed at 25% of the distance between the tip of the head of the fibula and the tip of the lateral malleolus.

In order to measure the maximum voluntary contraction values from the determined muscle groups, separate EMG measurements will be performed with 3 repetitions of maximal contraction of 5 seconds, with a resting period of 30 seconds between each of them. As a result of these measurements, the average of these 3 repetitions performed at the maximum activation level for each muscle of the individuals will be taken. Afterward, surface EMG measurements will be taken from the same muscle groups for 10 seconds during the foot shortening exercises while breathing and without breathing. According to the maximum voluntary contraction for each muscle, the muscle activation rates will be determined during the foot shortening exercises with and without breathing [activity muscle activation amount / Maximal voluntary contraction * 100 (% Maximum voluntary contraction)]. The sampling rate of the EMG signal will be set to 1000 Hz. A 20 Hz Butterworth High-Pass filter will be applied to all EMG recordings and RMS 100 ms will be selected and filtered for smoothing. Measured data will be analyzed using Noraxon MyoResearch XP software (version 1.08; Noraxon Inc, Scottsdale, AZ).

ELIGIBILITY:
Inclusion Criteria:

* age between 18-25 years
* having bilateral pes planus according to Navicular Drop Test

Exclusion Criteria:

* were having rigid pes planus, hallux valgus, hallux rigidus, epin calcanei, systemic, neurological, or orthopedic problems that can affect the lower extremity
* inflammatory arthritis; foot ankle surgery; diabetes; or toe deformities, such as claw toe, or hammertoe,

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2021-10-05 (Actual); Primary Completion 2021-12-10 (Actual); Study Completion 2022-10-20 (Actual)

PRIMARY OUTCOMES:
Measurement of the activity of the Abductor Hallucis Longus, Tibialis Anterior or, Peroneus Longus | 30 min
  Muscle activity will be measured by surface electromyography. Measurment of activity will be done in three condition. Firstly maximum contraction, secondly on standing condition maximum contraction muscle activity will be measured. Last condition is on standing with restiratory exercises maximum contraction of muscles will be measured. Consequently all parameters will be compared.

CONTACTS AND LOCATIONS:
Overall Officials: Tezel Şahan, pHD, Study Director — University of Health science
Locations (1):
- Tezel Yıldırım Şahan, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Choi JH, Cynn HS, Yi CH, Yoon TL, Baik SM. Effect of Isometric Hip Abduction on Foot and Ankle Muscle Activity and Medial Longitudinal Arch During Short-Foot Exercise in Individuals With Pes Planus. J Sport Rehabil. 2020 Jul 27;30(3):368-374. doi: 10.1123/jsr.2019-0310. PMID 32717719
- [Background] Unver B, Erdem EU, Akbas E. Effects of Short-Foot Exercises on Foot Posture, Pain, Disability, and Plantar Pressure in Pes Planus. J Sport Rehabil. 2019 Oct 18;29(4):436-440. doi: 10.1123/jsr.2018-0363. Print 2020 May 1. PMID 30860412
- [Background] Jung DY, Koh EK, Kwon OY. Effect of foot orthoses and short-foot exercise on the cross-sectional area of the abductor hallucis muscle in subjects with pes planus: a randomized controlled trial. J Back Musculoskelet Rehabil. 2011;24(4):225-31. doi: 10.3233/BMR-2011-0299. PMID 22142711